CLINICAL TRIAL: NCT05549856
Title: Official Title: Dry Suction Technique Versus Wet Suction Technique of Endoscopic Ultrasound-Guided Fine-needle Biopsy for Diagnosis of Solid Pancreatic Lesions: A Randomized Controlled Non-Inferiority Trial
Brief Title: Comparision of EUS-FNB Techniques for Diagnose of Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEC-2022-335
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Solid Pancreatic Lesions; EUS-FNB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry suction group (Experimental): 22G Franseen needle biopsy with dry suction technique(The puncture needle be filled with air)
  Interventions: Procedure: Dry suction
- Wet suction group (Active Comparator): 22G Franseen needle biopsy with wet suction(The puncture needle be filled with saline before sugry)
  Interventions: Procedure: Wet suction

INTERVENTIONS:
Procedure: Wet suction — The pancreatic solid lesions will be puncture with the 22G Acquire needle (Boston Scientific Corporation, Marlborough, MA, USA). Before puncturing the lesion, flush the needle with 5ml saline, then use a 10 ml syringe in order to replacing the column of air with fluid. After puncture, monitoring the puncture needle under US guidance in real time, the needle was moved back and forth about 10-20 times within the lesion using a fanning technique.
  Arms: Wet suction group
Procedure: Dry suction — The pancreatic solid lesions will be puncture with the 22G Acquire needle (Boston Scientific Corporation, Marlborough, MA, USA). The stylet is removed and a 10 ml air-filled pre-vacuum syringe is attached. After puncture, monitoring the puncture needle under US guidance in real time, the needle was moved back and forth about 10-20 times within the lesion using a fanning technique.
  Arms: Dry suction group

SUMMARY:
Studies have shown that the wet-suction technique in EUS-FNA generates better histological diagnostic accuracy and specimen quality than the dry-suction technique. However, studies on wet suction on the diagnostic accuracy of EUS-FNB is small and the conclusions are controversial. Besides, the optional numeber of passes for EUS-FNB has not been determined.

DETAILED DESCRIPTION:
The investigators aimed to design a large multicenter randomized trial to compare the diagnostic accuracy and the optimal number of passes required for EUS-FNB in solid pancreatic lesions using 22G Franseen under wet aspiration versus standard aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years;
* Patients with solid pancreatic lesions evidenced by CT or MRI who do not have a histopathological diagnosis.
* Plan to receive EUS-FNB.
* Able to obtained informed consent.

Exclusion Criteria:

* Had expected difficulty of endoscope insertion
* That no lesion in the pancreas is identified by EUS
* Use of anticoagulants/antiplatelet drugs that cannot be discontinued.
* Had a bleeding tendency, defined as an international normalized ratio of the prothrombin time >1.5 or a platelet count <50,000 cells/mL
* Other medical conditions that render the patient an unsuitable candidate for EUS-FNB.
* Vulnerable groups such as pregnant women or patients with mental disorders;
* Patients unable to understand and/or read the consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 12 months
  compare the rate of diagnostic accuracy of EUS- FNB using the two different suction techniques (dry suction and wet suction) in patients with solid pancreatic lesions.

SECONDARY OUTCOMES:
Samples tissue integrity | 12 months
  The tissue integrity on histological analysis was graded into 3 levels: Grade A, existing core tissue (defined as an architecturally intact piece of tissue with a long axis measuring at least 550 μm), which can clearlycharacterize the lesion, and is sufficient for diagnosis; Grade B, existing core fragments, which does not meet the criteria for architecturally intact histology, but can still yield a diagnosis based on cell morphology;and Grade C, no lesion tissue found, and a diagnosis cannot be made based on the sample.
Samples cellularity | 12 months
  The cellularity of the cytological specimens was graded into 3 levels as follows : Grade A, more than 4 clusters, with a minimum of 10 cells in each cluster; Grade B, approximately 2-4 clusters, with a minimum of 10 cells in each cluster; and Grade C, fewer than 2 clusters or no cellular smear.
the diagnostic in relation to the number of needle passes | 12 months
  the diagnostic accuracy of each needle
Time (minutes) of the procedures with dry suction and wet suction | 12 months
  Time of the procedure is defined by the time from flushing the needle with saline solution to the removal of the needle after the last pass.
Percentage of procedure related adverse events [Safety] | 24 months
  Intra-procedural and post-procedural adverse events in the 2 arms will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Li Yue, Doctor, Principal Investigator — Nanfang Hospital, Southern Medical University

REFERENCES:
- [Derived] Xu S, Guo J, Qin M, Meng Y, Xie F, Qiao W, Hu H, Peng P, Rownoak J, Heng S, Ung F, Ye Y, Wang J, Li W, Zou Y, Zou L, Huang S, Liu S, Wang J, Yao J, Li Y. Dry Suction Versus Wet Suction of Endoscopic Ultrasound-Guided Fine-Needle Biopsy for Diagnosis of Solid Pancreatic Lesions: A Multicenter Randomized Controlled Noninferiority Trial. Am J Gastroenterol. 2025 Nov 1;120(11):2529-2537. doi: 10.14309/ajg.0000000000003389. Epub 2025 Feb 27. PMID 40019152
- [Derived] Xu S, Wang J, Guo J, Xie F, Qiao W, Meng Y, Peng P, Hu H, Huang Y, Liu S, Qin M, Yao J, Li Y. Dry suction versus wet suction technique of endoscopic ultrasound-guided fine-needle biopsy for diagnosis of solid pancreatic lesions: study protocol of a multicenter randomized controlled non-inferiority trial. Trials. 2023 Dec 13;24(1):805. doi: 10.1186/s13063-023-07842-8. PMID 38093381